CLINICAL TRIAL: NCT03050528
Title: The ExACT Trial: The Effectiveness of Exercise Combined With Acceptance and Commitment Therapy Compared to a Standalone Supervised Exercise Intervention for Chronic Pain. A Randomised Controlled Trial
Brief Title: The Effectiveness of Exercise Combined With Acceptance and Commitment Therapy for Chronic Pain
Acronym: ExACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Mater Misericordiae University Hospital (Other); Health Research Board, Ireland (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/378/1864
Record Dates: First submitted 2017-02-06; First posted 2017-02-13 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain
Keywords: Acceptance and Commitment Therapy; Exercise; Psychology; Psychological therapy; Physiotherapy; Physical therapy
MeSH Terms: conditions — Chronic Pain; Motor Activity | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The academic Statistician (Dr Ricardo Segurado) and the Senior Researcher (Maire-Brid Casey) will be blind to group allocation. Dr Segurado will be responsible for data analysis. Máire-Bríd Casey will be responsible for data entry and will assist with data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Exercise and ACT treatment (Experimental): Participants will attend a weekly group-based multidisciplinary pain programme for a period of eight weeks. The programme will combine exercise with the psychological approach acceptance and commitment therapy (ACT).
  Interventions: Behavioral: Supervised Exercise; Behavioral: Acceptance and Commitment Therapy
- Standalone supervised exercise (Active Comparator): Participants will attend a weekly group-based supervised exercise class for a period of eight weeks.
  Interventions: Behavioral: Supervised Exercise

INTERVENTIONS:
Behavioral: Supervised Exercise — Participants will attend the weekly supervised exercise sessions for a period of eight weeks. The classes will be delivered to groups of up to ten participants and will be led by a physiotherapist. The classes will be one hour and thirty minutes in duration and will feature two components: education/advice and exercise. The education/advice sessions will cover topics such as pacing and goal setting and the physiotherapist will answer any queries from the participants in relation to physical activity over the course of the eight weeks. The exercise component will involve the provision of individualised exercises based on each participant's personal goals and the sessions will feature a combination of aerobic, stretching and strengthening exercise in a pool and a gym setting.
Behavioral: Acceptance and Commitment Therapy — Participants will attend weekly group psychology sessions for an eight-week period. Each session will be two hours in duration and will delivered by a Senior Psychologist trained in Acceptance and Commitment Therapy (ACT). The sessions will feature an ACT treatment process that is designed to promote psychological flexibility through various methods including acceptance and values awareness. The overall aim is to promote behaviour change, enhancing patient engagement in meaningful activities and reducing pain-avoidant behaviours. There is an emphasis on mindfulness, experiential learning and the use of metaphor which is unique to ACT.
  Arms: Combined Exercise and ACT treatment

SUMMARY:
The aim of this study is to evaluate the effectiveness of a combined Exercise and Acceptance and Commitment Therapy (ACT) programme, compared to a standalone supervised exercise intervention for patients with chronic pain. Chronic pain is a common problem, which can have a significant impact on quality of life. While there are many treatments available for chronic pain, research has shown that improvements are often modest and short-term.

Exercise therapy is known to be helpful for many chronic conditions and is recommended in clinical guidelines for the management of chronic pain. Acceptance and Commitment Therapy (ACT) is a form of psychological therapy, which focuses on improvement of function, rather than symptom reduction. There is an emphasis on psychological flexibility, values and mindfulness. This approach may be well suited to chronic pain, where symptoms can be beyond a person's control, but there is a need for further research, particularly with regards to combining ACT with a physical intervention.

This study will take place in a Dublin University hospital. Patients will be randomly allocated to a combined exercise and ACT treatment group or a standalone exercise group. Both groups will have weekly treatment for eight weeks and will be assessed before and after treatment, and again twelve weeks later. Questionnaires will be used to measure the effects of the treatment on the degree to which pain interferes with various aspects of daily life. Activity trackers will be worn to measure daily physical activity levels. A purposeful sample of participants from both groups will also be invited to participate in a qualitative study following treatment.

DETAILED DESCRIPTION:
This prospective, two-armed, parallel group, single-centre Randomised Controlled Trial (RCT) will assess the effectiveness of a combined Exercise and ACT programme, in comparison to a standalone supervised exercise intervention for chronic pain. One hundred and sixty patients aged 18 years and over, who have been diagnosed with a chronic pain condition by a medical doctor will be recruited to the trial. Participants will be individually randomised to one of two group interventions. The combined group will take part in eight, weekly psychology sessions based on the ACT approach, in addition to supervised exercise classes led by a physiotherapist. The control group will also attend eight, weekly supervised exercise classes but will not take part in ACT programme. All participants will be assessed at baseline, immediately post intervention and at twelve-week follow-up. The primary outcome will be pain interference at twelve-week follow-up, measured using the Brief Pain Inventory-Interference Scale. Secondary outcomes will include self-reported pain severity, pain related self-efficacy, quality of life, kinesiophobia, pain catastrophizing, pain acceptance, committed action, patient global impression of change, patient satisfaction with treatment, depression and anxiety. The number of investigations and pain related visits to healthcare professionals in the preceding three months will be recorded at baseline and twelve-week follow-up. Physical activity levels (average daily step count, distance travelled and active minutes) will be measured for all participants using Fitbit Zip activity trackers for one week prior to starting treatment and for the duration of the eight week intervention period. Participants will be invited to wear the activity trackers for one further week at the twelve-week follow-up time point.

Estimates of treatment effects at follow up time-points will be based on an intention-to-treat framework, implemented using a linear mixed effects model. A purposeful sample of participants will be invited to attend individual interviews and focus groups, twelve weeks following completion of the interventions. Semi-structured interviews will be conducted, with the aim of exploring the views of participants of both interventions in order to enhance understanding of how these types of interventions work.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and over who have been diagnosed with chronic pain by a medical doctor
* Presence of persistent pain of greater than 12 weeks
* Ability to provide informed consent
* Ability to communicate adequately in spoken and written english
* Score of ≥ 3 on pain interference subscale of the Brief Pain Inventory

Exclusion Criteria:

* Need for further diagnostic evaluation
* Presence of major medical or psychiatric disorder which would impede ability to participate with treatment
* Presence of active cancer or cancer related pain
* Unstable inflammatory condition e.g. rheumatoid arthritis or gout
* Surgical or pain interventional procedure (e.g. spinal cord stimulator, rhizotomy, intra-articular or epidural injection) during the last 3 months.
* Concurrent participation, or participation in the previous 3 months with any form of psychological therapy, physiotherapy or supervised exercise intervention
* Previous participation in any form of multidisciplinary pain management programme
* Presence of substance misuse
* Presence of any contraindication to participation in a gym or pool based exercise programme such as shortness of breath at rest, unstable diabetes or epilepsy, recent myocardial infarction, stroke, pulmonary embolism, asthma attack
* Weight > 125 kg or waist circumference > 50 inches (restriction die to pool evacuation equipment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change in pain interference measured with the Brief Pain Inventory - Interference scale | 12 week follow up (20 weeks from baseline assessment)
  The interference subscale of the Brief Pain Inventory is a seven item self-report questionnaire that measures the extent to which pain interferes with functions such as general activity, walking ability, normal work, mood, relations with people, enjoyment of life and sleep.

SECONDARY OUTCOMES:
Change in pain interference measured with the Brief Pain Inventory Interference Scale | immediately post intervention (8 weeks from baseline)
  The interference subscale of the Brief Pain Inventory is a seven item self-report questionnaire that measures the extent to which pain interferes with functions such as general activity, walking ability, normal work, mood, relations with people, enjoyment of life and sleep.
Change in pain severity measured with the Brief Pain Inventory (BPI) Composite pain score | immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  Pain Severity will be measured using the composite pain score of the BPI
Change in pain self efficacy measured with the Pain Self Efficacy Questionnaire (PSEQ) | Immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  The PSEQ is a ten item questionnaire which assesses an individual's confidence in their ability to perform a variety of activities or tasks despite pain.
Change in quality of life measured with the EQ-5D-5L | Immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  The EQ-5D-5L assesses quality of life in five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Change in fear of movement measured with the Tampa Scale for Kinesiophobia (TSK) | Immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  Fear of movement or re-injury has been reported to be a strong predictor of physical functioning and disability in chronic pain. The TSK is reported to be reliable and valid measure of fear of movement in individuals with chronic pain.
Change in pain catastrophising measured with the Pain Catastrophising Scale (PCS) | Immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  The PCS is a 13-item instrument designed to assess catastrophic thinking in relation to pain. The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness.
Change in pain acceptance measured with the Chronic Pain Acceptance Questionnaire (CPAQ - 8) | Immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  Pain acceptance is considered to be a treatment process variable and is regularly used in studies which feature ACT. The CPAQ-8 is a shortened version of the original 20-item CPAQ with two subscales; activity engagement and pain willingness.
Change in committed action measured with the Committed Action Questionnaire (CAQ-8) | Immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  Committed action is another treatment process variable which we propose to measure. The CAQ-8 is a shortened version of the original 18-item Committed Action Questionnaire which measures committed action in relation to commitment to valued goals.
Patient Global Impression of Change Scale (PGIC) | Immediately post intervention (8 weeks from baseline)
  The PGIC scale measures a patient's rating of overall improvement or lack thereof due to the intervention.
Patient satisfaction with treatment measured with a single question from the Client Satisfaction Questionnaire-8 | Immediately post intervention (8 weeks from baseline)
  Satisfaction with treatment will be measured using a single question from the Client Satisfaction questionnaire (CSQ-8) which is designed to measure satisfaction with services. The question will ask "In an overall, general sense, how satisfied are you with the service you have received?" and four potential responses will be provided (very satisfied, mostly satisfied, indifferent or mildly dissatisfied and quite dissatisfied). The percentages of participants endorsing each of the responses will be reported.
Change in symptoms of depression measured using the Patient Health Questionnaire-9 (PHQ-9) | Immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  Symptoms of depression will be assessed using the PHQ-9, which is a nine-item questionnaire generating scores ranging from 0 - 27.
Change in symptoms of anxiety measured with the General Anxiety Disorder-7 questionnaire (GAD-7) | Immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  The GAD-7 assesses symptoms of anxiety experienced during the last two weeks.
Change in self-reported healthcare utilisation | Immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  This questionnaire will collect data related to healthcare utilisation during the preceding three month period including GP visits, hospital consultant visits, visits to alternative health care practitioners, emergency department visits and number of nights of hospital in-patient stay.
Change in physical activity levels (average weekly step count, distance travelled and active minutes) | Immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  Average weekly step count, distance travelled and active minutes will be measured using a FitBit Zip activity tracker for one week prior to randomisation and for the duration of the eight week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maire-Brid Casey, BSc, MMT, Principal Investigator — University College Dublin
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Raftery MN, Ryan P, Normand C, Murphy AW, de la Harpe D, McGuire BE. The economic cost of chronic noncancer pain in Ireland: results from the PRIME study, part 2. J Pain. 2012 Feb;13(2):139-45. doi: 10.1016/j.jpain.2011.10.004. PMID 22300900
- [Background] Williams AC, Eccleston C, Morley S. Psychological therapies for the management of chronic pain (excluding headache) in adults. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD007407. doi: 10.1002/14651858.CD007407.pub3. PMID 23152245
- [Background] Veehof MM, Oskam MJ, Schreurs KMG, Bohlmeijer ET. Acceptance-based interventions for the treatment of chronic pain: a systematic review and meta-analysis. Pain. 2011 Mar;152(3):533-542. doi: 10.1016/j.pain.2010.11.002. Epub 2011 Jan 19. PMID 21251756
- [Background] Wetherell JL, Afari N, Rutledge T, Sorrell JT, Stoddard JA, Petkus AJ, Solomon BC, Lehman DH, Liu L, Lang AJ, Atkinson HJ. A randomized, controlled trial of acceptance and commitment therapy and cognitive-behavioral therapy for chronic pain. Pain. 2011 Sep;152(9):2098-2107. doi: 10.1016/j.pain.2011.05.016. Epub 2011 Jun 17. PMID 21683527
- [Derived] Casey MB, Smart KM, Segurado R, Hearty C, Gopal H, Lowry D, Flanagan D, McCracken L, Doody C. Exercise combined with Acceptance and Commitment Therapy compared with a standalone supervised exercise programme for adults with chronic pain: a randomised controlled trial. Pain. 2022 Jun 1;163(6):1158-1171. doi: 10.1097/j.pain.0000000000002487. Epub 2021 Sep 24. PMID 34913883
- [Derived] Casey MB, Smart K, Segurado R, Hearty C, Gopal H, Lowry D, Flanagan D, McCracken L, Doody C. Exercise combined with Acceptance and Commitment Therapy (ExACT) compared to a supervised exercise programme for adults with chronic pain: study protocol for a randomised controlled trial. Trials. 2018 Mar 22;19(1):194. doi: 10.1186/s13063-018-2543-5. PMID 29566744